CLINICAL TRIAL: NCT00844740
Title: Effect of Cinacalcet on the Long-term Treatment of Familial Hypophosphatemic Rickets
Brief Title: Calcimimetics in Hypophosphatemic Rickets
Acronym: CHR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08 09-152
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Familial Hypophosphatemic Rickets
Keywords: Familial hypophosphatemic rickets; Cinacalcet; hyperparathyroidism
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Hyperparathyroidism | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cinacalcet (Experimental): Stable patients with XLH already treated with Phosphate and calcitriol will add Cinacalcet to their treatment regimen. Sequential monitoring of blood and urine biochemical variables will follow, based on which adjustments to the doses of the 3 medications will be done.
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — Stable patients with XLH already treated with Phosphate and calcitriol will add Cinacalcet to their treatment regimen. Sequential monitoring of blood nand urine biochemical variables will follow, based on which adjustments to the doses of the 3 medications will be done.
  Other Names: Sensipar

SUMMARY:
Currently, large oral doses of phosphate and 1,25(OH)2D (calcitriol) are the standard treatment of patients with familial hypophosphatemic rickets (XLH). While this therapy is effective in healing the rickets, it is often limited by development of complications due to the high dose of medications required to achieve cure. Among them are the development of calcifications in the kidneys and secondary hyperparathyroidism (HPT) which in some patients may cause complications like high blood calcium level, high blood pressure and damage to the kidney. A drug to treat secondary hyperparathyroidism was just developed. In a short term study we found that it might help the treatment of XLH, by allowing the use of lower doses of the both phosphate and calcitriol. In the present study we will learn if indeed the addition of this new medicine (Cinacalcet) to the long-term treatment will allow the use of lower doses of both phosphate and calcitriol and consequently lower the risk of complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with XLH
2. Age 5-21 years old
3. From the Renal and Endocrinology Clinics who have been in a stable clinical, biochemical and radiological condition for the preceding 9 months
4. Who have not received Cinacalcet before

Exclusion Criteria:

1. Treatment with growth hormone
2. Inability to swallow pills.
3. An orthopedic surgery or braces in the past 9 months, or scheduled within 9 months of start.
4. Pregnancy
5. History of seizure disorder
6. Abnormal liver functions (which may change the drug's AUC)

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03-01 (Estimated); Primary Completion 2012-03-01 (Estimated); Study Completion 2012-03-01 (Estimated)

PRIMARY OUTCOMES:
doses of phosphate and calcitriol required to sustain goals of blood and urine chemistries | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States